CLINICAL TRIAL: NCT06232096
Title: A Phase Ⅰ/Ⅱ Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of MBS314 Injection in Patients With Relapsed/Refractory Multiple Myeloma.
Brief Title: A Study of MBS314 in Participants With Relapsed/Refractory Multiple Myeloma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBS314-CT101
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBS314 (Experimental)
  Interventions: Drug: MBS314 Injection

INTERVENTIONS:
Drug: MBS314 Injection — Phase Ia: The patients confirming to the eligibility criteria will be assigned to 1 of the 7 dose groups (0.03/0.09/0.3/0.9 mg ~ 0.3/1.5/9.0/60 mg, respectively) based on the sequence of inclusion. Each patient will receive MBS314 as per the schedule specified in the respective arms.
  Phase Ib/Ⅱ: Based on the results of Phase Ⅰa, 1 or 2 recommended doses will be selected for Phase Ⅰb. Recommended Phase II Dose (RP2D) will be selected for Phase Ⅱ.

SUMMARY:
This is a Phase I/Ⅱ, multicenter, open-label, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics(PD) and efficacy of a novel asymmetric trivalent tri-specific humanized antibody, MBS314, administered by intravenous (IV) infusion in participants with relapsed or refractory multiple myeloma. This entry-to-human study is divided in 2 parts: a dose escalation part (Phase Ⅰa) and an expansion part (Phase Ⅰb/Ⅱ).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol;
2. ≥18 years of age;
3. Documented diagnosis of multiple myeloma according to 2014 IMWG diagnostic criteria.
4. Phase Ⅰb/Ⅱ: At least one measurable disease: Serum monoclonal paraprotein (M-protein) ≥5 g/L or Urine M-protein ≥200 mg/24 hours or Serum immunoglobulin free-light chains (FLCs) ≥100 mg/L and abnormal kappa/lambda FLC ratio (<0.26 or >1.65)
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
6. Life expectancy ≥3 months.
7. Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

1. Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
2. Participants with known active infection within 14 days prior to the first MBS314.
3. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C (including HBsAg, HBcAb positive with abnormal hepatitis B virus DNA or hepatitis C virus RNA).
4. Previously received anti-myeloma treatment within the specified time frame prior to the first administration.
5. Live, attenuated vaccines within 28 days prior to the first infusion of MBS314, or expected to receive live, attenuated vaccines during the study period.
6. Major surgery within 28 days prior to the first infusion of MBS314, or expected to undergo major surgery during the study treatment.
7. Participants with a history of autoimmune diseases.
8. Known severe allergic reactions to other antibodies, or known allergies or hypersensitivity to any components of MBS314.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase Ia:Percentage of Participants with Adverse Events (AEs) . | From Baseline up to approximately 29 months
  Percentage of Participants with AEs and serious adverse events Assessed by NCI CTCAE v5.0.
Phase Ia:Incidence of Dose Limiting Toxicities (DLTs) | From Baseline up to 4 weeks
  DLTs:Incidence of Dose Limiting Toxicities
Phase Ia:Maximum Tolerated Dose (MTD) of MBS314 | Up to approximately 11 months
  MTD:Maximum Tolerated Dose
Phase Ia:Recommended Phase Ⅱ Dose (RP2D) of MBS314 | Up to approximately 29 months
  RP2D: Recommended Phase II Dose
Phase Ib/Ⅱ :Efficacy: Overall Response Rate (ORR) as Assessed by Independent Review Committee (IRC) | Up to approximately 4 years
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the International Myeloma Working Group (IMWG) response criteria assessed by the IRC.

SECONDARY OUTCOMES:
Efficacy: Stringent Complete Response (sCR) Rate | Up to approximately 4 year
  sCR rate is defined as the percentage of patients who achieve a stringent complete response (sCR) according to the IMWG response criteria.
Efficacy: Complete Response (CR) or Better Rate | Up to approximately 4 year
  CR or better rate is defined as the percentage of patients who achieve a complete response (CR) or better according to the IMWG response criteria.
Efficacy: Minimal Residual Disease (MRD) Negative Rate | Up to approximately 4 years
  Minimal Residual Disease (MRD) Negative Rate
Efficacy: Very Good Partial Response (VGPR) or Better Rate | Up to approximately 4 year
  VGPR or better rate is defined as the percentage of patients who achieve a VGPR or better according to the IMWG response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No